CLINICAL TRIAL: NCT05253404
Title: Laryngeal Mask Airway Facilitates a Safe and Smooth Emergence From Anesthesia in Patients Undergoing Craniotomy: A Prospective Randomized Controlled Study
Brief Title: Laryngeal Mask Airway Facilitates a Safe and Smooth Emergence From Anesthesia in Patients Undergoing Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei. Cheng-Fong, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202102115A3
Record Dates: First submitted 2022-02-08; First posted 2022-02-23 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Complications, Pulmonary
Keywords: Extubation; Laryngeal mask; Craniotomies

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will going general anesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthesia remove endotracheal tube (No Intervention): When craniotomy surgery was done, inhalation anesthestic sevoflurane level will control at MAC 2-3%, at the same time we perform suction secretions in endotracheal tube and oral cavity and give neostigmine 0.05-0.07 mg/kg and glycopyrrolate 0.01mg/kg via intravascular catheter. Removing endotracheal tube when spontaneously generating tidal volume of >4ml/kg, EtCO2<45mmHg, Train of four ratio >70-90%.
- Switching endotracheal tube to laryngeal mask (Experimental): When craniotomy surgery was done, inhalation anesthestic sevoflurane level will control at 2.63%-2.97%, we perform suction secretions in endotracheal tube and oral cavity, then switching endotracheal tube to laryngeal mask. Then we discontinue inhalation anesthestic sevoflurane and support oxygen at the rate of 6L/min. At the same time, give neostigmine 0.05-0.07 mg/kg and glycopyrrolate 0.01mg/kg via intravascular catheter. Removing endotracheal tube when sevofulrane at MAC 0.4, spontaneously generating tidal volume of >4ml/kg, EtCO2<45mmHg, Train of four ratio >70-90%.
  Interventions: Device: Ambu® AuraOnce™ Disposable Laryngeal Mask

INTERVENTIONS:
Device: Ambu® AuraOnce™ Disposable Laryngeal Mask — Switching endotracheal tube to laryngeal mask at sevoflurane 2.63-2.97%, Removing endotracheal tube when spontaneously generating tidal volume of >4ml/kg, EtCO2<45mmHg, Train of four ratio >70-90%.
  Arms: Switching endotracheal tube to laryngeal mask

SUMMARY:
Stabilizing hemodynamic and reducing pulmonary complications during extubation with switching endotracheal tube to laryngeal mask in craniotomies

DETAILED DESCRIPTION:
recruit ASA: 1-3, 20-65 years old undergoing neurosurgery under general anesthesia Excluded 1.Decline to participated 2.Difficult airway 3.Body Mass Index >30 4. Pregnant woman 5.Nothing Per Os <8hrs(case number:80).

General anesthesia Induction: 0.15-0.2 mg/kg cisatracurium or 0.6-1.2mg rocuronium , 1.5-2 mg/kg propofol, 1-2 mcg/kg Fentanyl. Endotracheal tube 6.5-7.5mm. Maintenance with sevoflurane 2- 3% FiO2:100%. Optimal muscle tension monitor. When surgery done, sevoflurane at 2.63-2.97%

Then randomly assigned two group Anesthesia group(control group) : Removed endotracheal tube at sevoflurane at 2-3% Switching group (intervention group): Intervention with endotracheal tube to laryngeal mask, and removing laryngeal mask at sevoflurane: 0.4MAC

ELIGIBILITY:
Inclusion Criteria:

* ASA: 1-3, 20-65 years old undergoing craniotomies under general anesthesia

Exclusion Criteria:

* Decline to participated
* Difficult airway
* Body Mass Index >30
* Pregnant woman
* Nothing Per Os <8hrs

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Hemodynamic | 30 minutes
  Blood pressure including systolic, diastolic and mean arterial pressure and heart rate during extubation
Pulmonary complications | 24 hours
  Rate of Participants with Cough, Bucking, Laryngospasm, Aspiration, Desaturation(SpO2%< 90%) and Need airway assist device(Nasal or oral airway)
Partial pressure of carbon dioxide in arterial blood | 20 mins
  Partial pressure of carbon dioxide in arterial blood five minutes before and after extubation

SECONDARY OUTCOMES:
Re-do surgery | 24 hours
  Number of Participants with Re-do neurosurgery within 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tai Chung, MD, Principal Investigator — Chang Gung Memorial Hospital; Cheng-Fong Wei, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Wei Cheng-Fong, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suppiah RK, Rajan S, Paul J, Kumar L. Respiratory and hemodynamic outcomes following exchange extubation with laryngeal mask airway as compared to traditional awake extubation. Anesth Essays Res. 2016 May-Aug;10(2):212-7. doi: 10.4103/0259-1162.174469. PMID 27212749
- [Background] Koga K, Asai T, Vaughan RS, Latto IP. Respiratory complications associated with tracheal extubation. Timing of tracheal extubation and use of the laryngeal mask during emergence from anaesthesia. Anaesthesia. 1998 Jun;53(6):540-4. doi: 10.1046/j.1365-2044.1998.00397.x. PMID 9709138
- [Background] Wong TH, Weber G, Abramowicz AE. Smooth Extubation and Smooth Emergence Techniques: A Narrative Review. Anesthesiol Res Pract. 2021 Jan 15;2021:8883257. doi: 10.1155/2021/8883257. eCollection 2021. PMID 33510786
- [Background] Juang J, Cordoba M, Ciaramella A, Xiao M, Goldfarb J, Bayter JE, Macias AA. Incidence of airway complications associated with deep extubation in adults. BMC Anesthesiol. 2020 Oct 29;20(1):274. doi: 10.1186/s12871-020-01191-8. PMID 33121440
- [Derived] Wei CF, Chung YT. Laryngeal mask airway facilitates a safe and smooth emergence from anesthesia in patients undergoing craniotomy: a prospective randomized controlled study. BMC Anesthesiol. 2023 Jan 17;23(1):29. doi: 10.1186/s12871-023-01972-x. PMID 36650435